CLINICAL TRIAL: NCT02991417
Title: Safety and Immunogenicity Study of a Clostridium Difficile Vaccine in Healthy Adult Volunteers
Brief Title: Oral Vaccination Against Clostridium Difficile Infection
Acronym: CDVAX
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Simon M. Cutting (Other)
Responsible Party: Sponsor-Investigator, Simon M. Cutting, Professor, Royal Holloway University
Organization: Royal Holloway University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDVAX
Record Dates: First submitted 2016-12-05; First posted 2016-12-13 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

ARMS (1):
- CDVAX (Experimental)
  Interventions: Biological: CDVAX

INTERVENTIONS:
Biological: CDVAX

SUMMARY:
This clinical study is conducted to assess the safety and immunogenicity of a Clostridium difficile vaccine (CDVAX) in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Male
3. Age: 18-50 years (limits included)
4. Body mass index within 18.5 and 29.9 kg/m²
5. Ability to read and comprehend study information
6. Non-smokers or light smokers (<4 cigarettes per day)
7. In good physical and mental health as determined by the following:

   1. Complete medical history
   2. Complete physical and neurological examination
   3. Vital signs including blood pressure, heart rate, respiratory rate, and temperature
   4. Standard 12-lead ECG
   5. Clinical laboratory (biochemistry, haematology and urinalysis) tests. Blood and urine samples may be drawn up to 3 weeks prior to the baseline visit of the study provided all data are available and evaluated prior to administration of study drug. Values of laboratory results outside normal reference ranges may be acceptable if the investigator considers that they do not compromise the safety of the subjects or the conduct of the study.
   6. Vital signs, clinical laboratory measurements, and ECG measurements may be repeated at the discretion of the investigator

Exclusion Criteria:

1. Evidence of C. difficile infection
2. Anti-C. difficile (Toxin A) immunoreactivity, suggesting previous C. difficile exposure
3. Diarrhoea, active or inactive inflammatory bowel disease, irritable colon syndrome, chronic abdominal pain or other chronic diarrhoea
4. History of malignancy within 5 years
5. History of anaphylaxis, asthma or severe vaccine or allergic drug reaction
6. Known or suspected history of immunodeficiency, active or inactive immune-mediated or inflammatory disease
7. Receipt of antibiotic therapy, immunosuppressants, or corticosteroids within the previous 30 days
8. Vaccination within the previous 30 days (except for influenza vaccination)
9. Blood or organ donation within the previous 60 days
10. Evidence of clinically significant psychiatric, gastrointestinal, neurologic, neuromuscular, hepatic, pulmonary, cardiovascular, or renal disease (as judged by the investigator)
11. Use of prescription medication or regular use of over-the-counter medicines or herbal or dietary supplements. Acetaminophen/paracetamol may be used intermittently as needed for pain
12. History or current evidence of abuse of any drug substance, licit or illicit, including alcohol; a positive urine screen for drugs of abuse
13. Positive hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg) or positive human immunodeficiency virus (HIV)-1/2 antibodies
14. Participation in any other investigational drug or device study within 60 days prior to the first study drug administration
15. Relatives of, or staff directly reporting to the principal investigator
16. Vulnerable subjects

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | First treatment up to end of treatment + 28 days (70 days after treatment start)
  Measured by routine physical and laboratory evaluations, adverse event monitoring, ECG and neurological examination

SECONDARY OUTCOMES:
Evaluation of specific mucosal and systemic immunity | First treatment up to end of treatment + 14 days (56 days after starting study drug)
  Measured by specific secretory IgA, serum IgA and serum IgG